CLINICAL TRIAL: NCT06324500
Title: Prognostic Role of Bowel Ultrasound Scan in Children Affected by Acute Severe Colitis (ASC): A Prospective Multicenter Study From the Paediatric IBD Porto Group of ESPGHAN
Brief Title: Prognostic Role of Bowel Ultrasound Scan in Children Affected by Acute Severe Colitis
Status: Recruiting | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Paolo Lionetti, Full Professor, Head of Gastroenterology, Principal Investigator, Meyer Children's Hospital IRCCS
Other Study IDs: ASC-US
Record Dates: First submitted 2024-02-23; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Acute Severe Colitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ASC is a life-threatening medical emergency. The lack of a timely intervention has shown to be associated with a mortality rate higher than 20% in adults, whereas a prompt targeted therapy has displayed a decrease of the aforementioned rate to 1%. Therefore, the identification of predictors of poor outcome trough an objective tool may provide crucial help to individualize the timing of second line treatment initiation. At the state of the art, PUCAI represents the only validated tool to appraise the risk of first-line treatment failure and there is a lack of objective methods with a prognostic value in ASC.

BUS has proven to be a reliable tool in assessing disease activity in children with UC and it has also shown statistically significant correlation with endoscopic features of disease activity. Given the literature suggesting a role for BUS in severe UC and the results from our retrospective study we aim to validate our findings trough a prospective assessment of the potential prognostic role of BUS in ASC.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged < 18 years hospitalized for ASC with diagnosis of UC established by the presence of accepted clinical, radiologic, endoscopic, and histologic criteria

Exclusion Criteria:

* Patients with infectious colitis;
* Patients undergoing treatment with anti-TNF alpha agents;
* Patients already enrolled during the study period for a previous ASC attack;

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged < 18 years hospitalized for ASC with diagnosis of UC established by the presence of accepted clinical, radiologic, endoscopic, and histologic criteria
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2025-03-02 (Estimated); Study Completion 2025-05-02 (Estimated)

PRIMARY OUTCOMES:
Colonic wall thickness of BUS (bowel ultrasound) parameter to predict the failure of first line treatment | Within 48 hours from i.v. steroid treatment initiation
  Investigation of the ability of BUS (bowel ultrasound) parameters, such as Colonic wall thickness (CWT) measured in mm, assessed within 48 hours from i.v. steroid treatment initiation, to predict the failure of first line treatment (defined according to the latest ESPGHAN guidelines).
  CWT will be measured from the edge of the outer wall to the inner echogenic lumen, containing air, or to the central echogenic mucosal stripe. CWT will be assessed as follows: two measurement through longitudinal plain and two through tranverse plain will be performed and the mean value (the sum of each measurement divided for 4) will be taken into account
Color and power Doppler vascularization of BUS (bowel ultrasound) parameter to predict the failure of first line treatment | Within 48 hours from i.v. steroid treatment initiation
  Colonic wall vascularization will be assessed according to the Limberg score to identify two subgroups: 1) increased vascularization (Limberg score 3-4); 2) normal colonic wall flow (Limberg Score 0-2). Such classification will be used, measured within the first 48 hours from i.v. steroid initiation, to predict failure of first line treatment (according to the latest ESPGHAN guidelines)
Mesenteric lymph nodes BUS (bowel ultrasound) parameter | Within 48 hours from i.v. steroid treatment initiation
  Presence of enlarged mesenteric lymph nodes, defined by short axis > 5 mm it will be assessed within 48 hours from i.v. steroid treatment initiation, to predict the failure of first line treatment (defined according to the latest ESPGHAN guidelines)

SECONDARY OUTCOMES:
evaluation of the prognostic value of the ultrasound parameters | Within 48 hours from second-line therapy initiation
  evaluation of the prognostic value of the ultrasound parameters in predicting the possible failure of second-line therapy and therefore the need to carry out colectomy surgery

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Lionetti, MD, Principal Investigator — Meyer Children's Hospital IRCCS
Locations (4):
- Italy (3):
  - Meyer Children's Hospital IRCCS, Florence, Firenze
  - Ospedale Maggiore, Bologna
  - IRCCS Materno Infantile Burlo Garofolo, Trieste
- CMED Centro Médico-Quirúrgico de Enfermedades Digestivas, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No